CLINICAL TRIAL: NCT03551626
Title: COMBI-APlus: Open-label, Phase IIIb Study of Dabrafenib in COMBInation With Trametinib in the Adjuvant Treatment of Stage III BRAF V600 Mutation-positive Melanoma After Complete Resection to Evaluate the Impact on Pyrexia Related Outcomes of an Adapted Pyrexia AE-management Algorithm (Plus)
Brief Title: Study of Dabrafenib+Trametinib in the Adjuvant Treatment of Stage III BRAF V600+ Melanoma After Complete Resection to Evaluate the Impact on Pyrexia Related Outcomes
Acronym: COMBI-APlus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDRB436F2410; 2018-000168-27 (EudraCT Number)
Record Dates: First submitted 2018-04-30; First posted 2018-06-11 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Malignant Melanoma
Keywords: dabrafenib; trametinib; adjuvant; Stage III melanoma; combination treatment; pyrexia
MeSH Terms: conditions — Melanoma; Fever | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib and trametinib combination therapy (Experimental): Subjects received dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) orally for up to 12 months.
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Supplied as dabrafenib 50 mg and 75 mg capsules for oral administration
  Other Names: DRB436
Drug: Trametinib — Supplied as trametinib 0.5mg, and 2.0mg tablets for oral administration
  Other Names: TMT212

SUMMARY:
The main purpose of this study was to evaluate the impact on pyrexia-related outcomes of an adapted pyrexia adverse event (AE)-management algorithm, as well as safety, efficacy and health-related outcomes.

DETAILED DESCRIPTION:
This was an open-label Phase IIIb study of dabrafenib in combination with trametinib in the adjuvant treatment of melanoma after complete resection. Patients with completely resected, histologically confirmed, BRAF V600E/K mutation-positive, high-risk cutaneous melanoma were screened for eligibility.

This study consisted of two periods:

1. Treatment Period - patients received up to 12 months of dabrafenib (150 mg twice daily) and trametinib (2 mg once daily). In the adapted pyrexia management algorithm, dabrafenib and trametinib were interrupted promptly at the onset of pyrexia (≥38°C) and were restarted upon the improvement of symptoms at the same dose if patients remained symptom free (temperature <38°C) for at least 24 hours. In addition, dabrafenib and trametinib could be interrupted in the presence of pyrexia syndrome (i.e. chills, rigours, night sweats, or influenza-like symptoms) without documented temperature ≥38°C for cases of suspected recurrent pyrexia, at the investigators' discretion.
2. Follow-up Period - patients were followed for disease relapse through 24 months from first dose date. Moreover, patients were followed for overall survival through withdrawal, lost to follow-up, death, or the end of study, whichever occurs first. The follow-up period started once treatment was completed or treatment was prematurely discontinued.

ELIGIBILITY:
Key Inclusion Criteria:

* Completely resected histologically confirmed cutaneous melanoma stage IIIA (LN metastasis >1 mm), IIIB, IIIC, IIID [AJCC (ed 8)] no more than 12 weeks, from last surgery, before Day 1

  1. Subjects presenting with initial resectable lymph node recurrence after a diagnosis of Stage I or II melanoma were eligible.
  2. Subjects who had previously had Stage III melanoma at any time were not eligible.
  3. Recovered from definitive surgery (e.g. no uncontrolled wound infections or indwelling drains).
* V600E/K mutation positive using a validated local test
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1

Key Exclusion Criteria:

* Uveal or mucosal melanoma
* Evidence of metastatic disease including unresectable in-transit metastasis
* Received any prior adjuvant or neoadjuvant treatment, including but not limited to chemotherapy, checkpoint inhibitors, targeted therapy [e.g., BRAF and/or MEK inhibitors], biologic therapy, vaccine therapy, investigational treatment, or radiotherapy for melanoma
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and had not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers and any completely resected carcinoma in situ
* History or current evidence of cardiovascular risk
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (95):
- Argentina (3):
  - Novartis Investigative Site, Rosario, Sante Fe
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Australia (2):
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Cairns
- Brazil (3):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (8):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Czechia (8):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (20):
  - Novartis Investigative Site, Pierre-Bénite, Cedex 02
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Rennes, Ille Et Vilaine
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lorient
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (12):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Antella - Bagno A Ripoli, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Napoli
- Japan (2):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Vilnius, Lithuania
- Norway (2):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Oslo
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Porto, Portugal
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Moscow Region Istra Village
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Saint Petersburg
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- Novartis Investigative Site, Ljubljana, Slovenia
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
- Novartis Investigative Site, Izmir, Turkey (Türkiye)
- United Kingdom (7):
  - Novartis Investigative Site, Bristol, Avon
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Atkinson V, Robert C, Grob JJ, Gogas H, Dutriaux C, Demidov L, Gupta A, Menzies AM, Ryll B, Miranda F, Banerjee H, Lau M, Del Vecchio M. Improved pyrexia-related outcomes associated with an adapted pyrexia adverse event management algorithm in patients treated with adjuvant dabrafenib plus trametinib: Primary results of COMBI-APlus. Eur J Cancer. 2022 Mar;163:79-87. doi: 10.1016/j.ejca.2021.12.015. Epub 2022 Jan 14. PMID 35042070
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients in this study were enrolled at 103 centers across 23 countries
Pre-assignment Details: A total of 748 patients were screened. Of the screened patients, 552 patients were treated.
Groups:
- Dabrafenib+Trametinib: Subjects received dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) orally for up to 12 months.
Period: Overall Study
Arm/Group | Dabrafenib+Trametinib
Started | 552
Completed | 425
Not Completed | 127
Not completed — Adverse Event | 88
Not completed — Disease relapse | 18
Not completed — Withdrawal of informed consent | 6
Not completed — Patient decision | 5
Not completed — Physician Decision | 4
Not completed — Lost to Follow-up | 3
Not completed — Pregnancy | 1
Not completed — Protocol deviation | 1
Not completed — Technical problems | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255
  Male | 297
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 377
  Asian | 3
  Missing | 172

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of Pyrexia Related Events
Description: The composite rate of pyrexia related events was calculated as the total number of participants experiencing at least one of the three components of the composite endpoint (i.e., grade 3/4 pyrexia, hospitalization due to pyrexia, or permanent treatment discontinuation due to pyrexia), divided by the total number of participants treated in the study and multiplied by 100. Pyrexia is defined as fever ≥ 38 °C.
  Pyrexia events were graded by the investigator using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Life-threatening) and Grade 5 (Death)
Time Frame: Baseline up to 12 months
Population: All subjects who received at least one dose of any study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Percentage of participants | 7.6 [5.5 to 10.1]

2. Secondary Outcome: Relapse Free Survival (RFS) Rate
Description: RFS is defined as the time from the date of first dose of the study treatment to the date of the first documented disease recurrence or death due to any cause whichever comes first. Treatment emergent malignancies other than second melanomas were not considered as events.
  RFS rate is the estimated percent probability that a patient will remain event-free up to the specified time point. RFS rate was obtained from the Kaplan-Meier survival estimates. RFS was censored if no RFS event was observed before the first to occur between: (i) the analysis cut-off date, and (ii) the date when a new anti-cancer therapy is started. The censoring date was the date of the last adequate tumor assessment prior to data cut-off date/start of new anti-cancer therapy date.
Time Frame: At 12 and 24 months
Population: All subjects who received at least one dose of any study treatment
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Percent probability
  12 months | 91.7 [89.0 to 93.8]
  24 months | 57.5 [48.9 to 65.2]

3. Secondary Outcome: Overall Survival (OS) Rate
Description: OS is defined as the time from date of the first dose of study medication to date of death due to any cause, whichever comes first. If a patient was not known to have died, then OS rate is the estimated probability that a patient will remain event-free up to the specified time point. OS rate was obtained from the Kaplan-Meier survival estimates. OS was censored at the last contact date when the patient was known to be alive (on or before the cut-off date).
Time Frame: At 12 and 24 months
Population: All subjects who received at least one dose of any study treatment
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Percent probability
  12 months | 99.1 [97.8 to 99.6]
  24 months | 92.6 [90.0 to 94.5]

4. Secondary Outcome: Percentage of Participants Who Required Management of Pyrexia
Description: Percentage of patients who experienced pyrexia and required intervention including hospitalizations, concomitant medications, and study treatment modifications (dose reductions, permanent discontinuations and/or interruptions) due to pyrexia. Pyrexia is defined as fever ≥ 38 °C
Time Frame: Baseline up to 12 months
Population: All subjects who received at least one dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Participants
  Hospitalizations due to pyrexia | 24
  Concomitant medications due to pyrexia | 210
  Permanent discontinuation of dabrafenib and trametinib (both drugs together) due to pyrexia | 13
  Reduction of dabrafenib and trametinib (both drugs together) due to pyrexia | 29
  Interruption of dabrafenib and trametinib (both drugs together) due to pyrexia | 339

5. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Treatment Due to Any Adverse Event (AE)
Description: Percentage of participants who permanently discontinued treatment due to any AE during treatment. An AE is any untoward medical occurrence (e.g., any unfavorable and unintended sign, symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study.
Time Frame: Baseline up to 12 months
Population: All subjects who received at least one dose of any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Participants | 87

6. Secondary Outcome: Change From Baseline in Subject-reported Quality of Life (QoL) Assessed by Functional Assessment Cancer Therapy - Melanoma Subscale Score (FACT-M MS)
Description: The FACT-M is a questionnaire that assesses participant health-related quality of life. It includes a melanoma specific (FACT-M MS) subscale that consists in 16 items related to signs, symptoms, physical/social activities most relevant to participants with advanced-stage melanoma. Each item ranges from 0 (not at all) to 4 (very much). FACT-M MS score ranges from 0 to 64, with higher score indicating better quality of life. If a patient discontinued the study treatment at Month 1 or Month 2, then the follow-up assessments started at Month 3 follow-up and continued until Month 24 follow-up or at withdrawal, lost to follow-up, death, or end of study. If a patient discontinued the study treatment from Month 3 through Month 5, the follow-up assessments started at Month 6 follow-up. If a patient discontinued from Month 6 through Month 11, the follow-up assessments started from Month 12 follow-up. For patients who completed treatment, the follow-up assessments started from Month 15 follow-up
Time Frame: Baseline up to 24 months
Population: All subjects who received at least one dose of any study treatment. Number analyzed represents participants with data available at the specified data points
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Score on a scale
  Month 1: number analyzed (Participants) | 463
  Month 1 | -2.46 (5.488)
  Month 2: number analyzed (Participants) | 449
  Month 2 | -2.42 (4.892)
  Month 3: number analyzed (Participants) | 438
  Month 3 | -2.26 (4.789)
  Month 4: number analyzed (Participants) | 421
  Month 4 | -2.34 (5.297)
  Month 5: number analyzed (Participants) | 426
  Month 5 | -2.03 (5.278)
  Month 6: number analyzed (Participants) | 414
  Month 6 | -2.19 (5.494)
  Month 7: number analyzed (Participants) | 405
  Month 7 | -2.39 (5.873)
  Month 8: number analyzed (Participants) | 387
  Month 8 | -2.32 (5.609)
  Month 9: number analyzed (Participants) | 361
  Month 9 | -2.06 (5.534)
  Month 10: number analyzed (Participants) | 338
  Month 10 | -2.15 (5.743)
  Month 11: number analyzed (Participants) | 326
  Month 11 | -2.05 (5.578)
  Month 12: number analyzed (Participants) | 316
  Month 12 | -1.96 (5.757)
  End of treatment: number analyzed (Participants) | 72
  End of treatment | -3.36 (5.944)
  Follow-up Month 3: number analyzed (Participants) | 7
  Follow-up Month 3 | 2.43 (4.685)
  Follow-up Month 6: number analyzed (Participants) | 27
  Follow-up Month 6 | -0.33 (4.915)
  Follow-up Month 12: number analyzed (Participants) | 38
  Follow-up Month 12 | -1.71 (5.671)
  Follow-up Month 15: number analyzed (Participants) | 260
  Follow-up Month 15 | -0.60 (6.018)
  Follow-up Month 18: number analyzed (Participants) | 269
  Follow-up Month 18 | -0.09 (4.948)
  Follow-up Month 24: number analyzed (Participants) | 271
  Follow-up Month 24 | -0.75 (5.406)

7. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from date of first administration of study treatment to 30 days after date of last administration of any study treatment (dabrafenib or trametinib).
  Post-treatment follow-up deaths were collected after the on-treatment period. All deaths refer to the sum of on-treatment and post-treatment follow-up deaths
Time Frame: On-treatment: from first study treatment to 30 days after last dose of study treatment, up to 13 months. Post-treatment: From day 31 after last study treatment up to approximately 39 months
Population: All subjects who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib+Trametinib
Number analyzed (Participants) | 552
Participants
  On-treatment deaths | 1
  Post-treatment follow-up deaths: number analyzed (Participants) | 537
  Post-treatment follow-up deaths | 47
  All deaths | 48

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of first administration of study treatment to 30 days after date of last actual administration of any study treatment (dabrafenib or trametinib), up to approximately 13 months. Deahs were collected in the post-treatment follow-up period from 31 days after last dose of study treatment until the end of the study, up to approximately 39 months
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment (on-treatment period). Deaths in the post treatment follow-up are not considered Adverse Events. The total number at risk in the post-treatment period includes patients that entered the post-treatment follow-up period.
Groups:
- Dabrafenib+Trametinib (On-treatment): AEs during on-treatment period (up to 30 days post-treatment)
- Dabrafenib+Trametinib (Post-treatment Follow-up): Deaths collected in the post-treatment follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Dabrafenib+Trametinib (On-treatment) | Dabrafenib+Trametinib (Post-treatment Follow-up)
All-Cause Mortality (participants affected / at risk) | 1/552 | 47/537
Serious Adverse Events (participants affected / at risk) | 121/552 | 0/0
Other Adverse Events (participants affected / at risk) | 526/552 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib+Trametinib (On-treatment) (N=552) | Dabrafenib+Trametinib (Post-treatment Follow-up) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | NA
Atrial fibrillation (Cardiac disorders) | 3 | NA
Left ventricular dysfunction (Cardiac disorders) | 2 | NA
Angina pectoris (Cardiac disorders) | 1 | NA
Cardiac failure (Cardiac disorders) | 1 | NA
Detachment of retinal pigment epithelium (Eye disorders) | 1 | NA
Retinal vein occlusion (Eye disorders) | 1 | NA
Scleritis (Eye disorders) | 1 | NA
Uveitis (Eye disorders) | 1 | NA
Abdominal discomfort (Gastrointestinal disorders) | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 1 | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | NA
Diarrhoea (Gastrointestinal disorders) | 1 | NA
Haematemesis (Gastrointestinal disorders) | 1 | NA
Nausea (Gastrointestinal disorders) | 1 | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | NA
Vomiting (Gastrointestinal disorders) | 1 | NA
Pyrexia (General disorders) | 28 | NA
Influenza like illness (General disorders) | 3 | NA
Chills (General disorders) | 2 | NA
Chest pain (General disorders) | 1 | NA
Fatigue (General disorders) | 1 | NA
Granuloma (General disorders) | 1 | NA
Hyperthermia (General disorders) | 1 | NA
Cholestasis (Hepatobiliary disorders) | 1 | NA
Hepatotoxicity (Hepatobiliary disorders) | 1 | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | NA
Cellulitis (Infections and infestations) | 5 | NA
Erysipelas (Infections and infestations) | 3 | NA
Pneumonia legionella (Infections and infestations) | 2 | NA
Appendicitis (Infections and infestations) | 1 | NA
Bacterial infection (Infections and infestations) | 1 | NA
Complicated appendicitis (Infections and infestations) | 1 | NA
Groin infection (Infections and infestations) | 1 | NA
Infection (Infections and infestations) | 1 | NA
Lower respiratory tract infection (Infections and infestations) | 1 | NA
Peritonitis (Infections and infestations) | 1 | NA
Pneumonia (Infections and infestations) | 1 | NA
Pneumonia aspiration (Infections and infestations) | 1 | NA
Prostate infection (Infections and infestations) | 1 | NA
Sepsis (Infections and infestations) | 1 | NA
Soft tissue infection (Infections and infestations) | 1 | NA
Systemic candida (Infections and infestations) | 1 | NA
Seroma (Injury, poisoning and procedural complications) | 1 | NA
Ejection fraction decreased (Investigations) | 19 | NA
Alanine aminotransferase increased (Investigations) | 1 | NA
Aspartate aminotransferase increased (Investigations) | 1 | NA
General physical condition abnormal (Investigations) | 1 | NA
Hepatic enzyme increased (Investigations) | 1 | NA
Lipase increased (Investigations) | 1 | NA
Lymphocyte morphology abnormal (Investigations) | 1 | NA
Neutrophil count decreased (Investigations) | 1 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | NA
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Cerebrovascular accident (Nervous system disorders) | 1 | NA
Focal dyscognitive seizures (Nervous system disorders) | 1 | NA
Headache (Nervous system disorders) | 1 | NA
Loss of consciousness (Nervous system disorders) | 1 | NA
Multiple sclerosis (Nervous system disorders) | 1 | NA
Polyneuropathy (Nervous system disorders) | 1 | NA
Presyncope (Nervous system disorders) | 1 | NA
Radicular pain (Nervous system disorders) | 1 | NA
Major depression (Psychiatric disorders) | 1 | NA
Nephrolithiasis (Renal and urinary disorders) | 2 | NA
Haematuria (Renal and urinary disorders) | 1 | NA
Renal colic (Renal and urinary disorders) | 1 | NA
Renal failure (Renal and urinary disorders) | 1 | NA
Urinary retention (Renal and urinary disorders) | 1 | NA
Ovarian cyst (Reproductive system and breast disorders) | 1 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Rash (Skin and subcutaneous tissue disorders) | 2 | NA
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | NA
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | NA
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | NA
Skin mass (Skin and subcutaneous tissue disorders) | 1 | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | NA
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 | NA
Lymphoedema (Vascular disorders) | 1 | NA
Venous thrombosis (Vascular disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib+Trametinib (On-treatment) (N=552) | Dabrafenib+Trametinib (Post-treatment Follow-up) (N=0)
Neutropenia (Blood and lymphatic system disorders) | 44 | NA
Abdominal pain (Gastrointestinal disorders) | 44 | NA
Abdominal pain upper (Gastrointestinal disorders) | 30 | NA
Constipation (Gastrointestinal disorders) | 46 | NA
Diarrhoea (Gastrointestinal disorders) | 149 | NA
Nausea (Gastrointestinal disorders) | 128 | NA
Vomiting (Gastrointestinal disorders) | 84 | NA
Chills (General disorders) | 146 | NA
Fatigue (General disorders) | 142 | NA
Influenza like illness (General disorders) | 65 | NA
Oedema peripheral (General disorders) | 66 | NA
Pain (General disorders) | 28 | NA
Asthenia (General disorders) | 131 | NA
Pyrexia (General disorders) | 374 | NA
Alanine aminotransferase increased (Investigations) | 75 | NA
Amylase increased (Investigations) | 35 | NA
Aspartate aminotransferase increased (Investigations) | 74 | NA
Blood alkaline phosphatase increased (Investigations) | 37 | NA
Blood creatine phosphokinase increased (Investigations) | 168 | NA
Lipase increased (Investigations) | 72 | NA
Decreased appetite (Metabolism and nutrition disorders) | 38 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 38 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 116 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 39 | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 42 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 85 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 | NA
Dizziness (Nervous system disorders) | 31 | NA
Headache (Nervous system disorders) | 174 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 79 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 33 | NA
Erythema (Skin and subcutaneous tissue disorders) | 38 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 29 | NA
Rash (Skin and subcutaneous tissue disorders) | 116 | NA
Hypertension (Vascular disorders) | 41 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03551626/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03551626/SAP_001.pdf